CLINICAL TRIAL: NCT07253909
Title: Investigation of Factors Determining Upper Extremity Function in Patients With Reduced Ejection Fraction Heart Failure and Cardiac Implantable Electronic Devices
Brief Title: Upper Extremity Function in Patients With Reduced Ejection Fraction Heart Failure and Cardiac Implantable Electronic Devices
Status: Enrolling by invitation | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aynur Demirel, PT, PhD, Assoc. Prof., Hacettepe University
Other Study IDs: FTREK25/74
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure; Implantable Cardioverter Defibrillator (ICD); Cardiac Resynchronisation Therapy (CRT); Reduced Ejection Fraction Heart Failure
Keywords: function; upper extremity; heart failure; Implantable cardioverter defibrillator (ICD); Cardiac Resynchronisation Therapy (CRT); Reduced ejection fraction heart failure
MeSH Terms: conditions — Heart Failure; Heart Failure, Systolic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Reduced Ejection Fraction Heart Failure and Cardiac Implantable Electronic Devices: Patients with Reduced Ejection Fraction Heart Failure and Cardiac Implantable Electronic Devices
  Interventions: Other: Not applicable- observational study

INTERVENTIONS:
Other: Not applicable- observational study — Not applicable- observational study

SUMMARY:
The aim of this study is to evaluate in detail the factors that determine upper extremity function, determine its effect on prognosis, hospital admission, hospitalization, and mortality, and examine the results according to the use of different implantable cardiac implantable electronic devices.

DETAILED DESCRIPTION:
In accordance with the inclusion and exclusion criteria appropriate to the purpose of the study, patients with a diagnosis of reduced ejection fraction heart failure and a cardiac implantable electronic device will be included. The demographic and clinical data of the individuals will be recorded. Their functional levels will be determined according to the New York Heart Association (NYHA) classification. Hand grip strength will be measured using a hand dynamometer, upper extremity anaerobic capacity will be assessed using a medicine ball throw test, upper extremity aerobic capacity will be evaluated using an arm ergometer test, and upper extremity functional exercise capacity will be assessed using the Unsupported Upper-limb Exercise Test (UULEX) and the Upper Limb Functional Test (ULIFT). Lower extremity functional capacity will be determined using the one-minute sit-to-stand test, and lower extremity performance will be determined using the 4-meter walk test. The Seattle Heart Failure Model will be used to estimate mortality risk and average life expectancy. Upper extremity functional status will be assessed using the Quick Disability of the Arm, Shoulder, and Hand Questionnaire, activities of daily living using the Katz Activities of Daily Living Scale, and quality of life using the Minnesota Quality of Life Scale. Comorbidity status will be determined using the Charlson Comorbidity Index.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years,
* Left ventricular ejection fraction ≤40%,
* Implanted cardiac defibrillator (ICD) or cardiac resynchronization therapy (CRT),
* Diagnosed with heart failure,
* No complications found during the last device check,
* Clinically stable for the past month, with any accompanying chronic diseases (such as hypertension, diabetes) under control, and willing to participate in the study.

Exclusion Criteria:

* Patients with neurological, orthopedic, or psychiatric disorders,
* History of shoulder surgery or shoulder injury,
* Individuals with cognitive or mental disorders that would prevent them from understanding the tests administered in the study, or patients who are unwilling to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study sample consists of patients with reduced ejection fraction heart failure who have a cardiac implantable electronic device, who meet the inclusion criteria, and who volunteer to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
upper extremity anaerobic capacity | one day
  Upper extremity anaerobic capacity will be assessed using the medicine ball throw test. Each patient will be asked to sit with one hand on their chest and throw a 2 kg medicine ball forward with the other hand. After the throw, the spot where the ball first touches the ground will be marked. Scores will be measured in centimeters, then the arithmetic mean will be calculated and recorded.
upper extremity aerobic capacity | one day
  Upper extremity aerobic capacity will be assessed using a arm ergometer test. The arm height of the ergometer will be set at shoulder level while seated. After the initial measurements are taken, the arm ergometer will be turned at a load of 0 watts and a speed of 60-75 rpm, and the load will be increased by 10 W every 2 minutes. The peak load reached by the patient will be recorded in watts.
Unsupported Upper-limb Exercise Test (UULEX) | one day
  The UULEX contain 8 horizontal levels. Each level is 84 cm wide and 8 cm high, with a distance of 15 cm between level centers. The lowest line corresponds to the participant's knee level. The participant holds a 0.2 kg plastic bar with their arms shoulder-width apart and moves it from the hips toward different levels. Each movement starts at the participant's hip joint and ends at the hip joint. After completing the first level for 2 minutes, the next levels are performed for 1 minute each. The bar is lifted up to 30 times per minute to the beat of a metronome. When participants reach their maximum height, the 0.2 kg bar is replaced with a 0.5 kg bar. They continue lifting to the maximum height with this weight. Then, the weight is increased by 0.5 kg every minute up to 2 kg. The time individuals can perform the test, the maximum weight they reach, and the level achieved will be recorded.
Upper Limb Functional Test (ULIFT) | one day
  The ULIFT is a performance test based on the Glittre test, developed to assess upper extremity functional capacity. ULIFT aims to objectively measure upper extremity function, endurance, and capacity for participation in activities of daily living, particularly through lifting movements and range of motion. Participants stand in front of shelves and, using one hand, carry three objects (weighing 1 kg each) from the top shelf (at shoulder height) to the bottom shelf (at waist height) and then from the bottom shelf to the floor; the objects are then returned to the bottom shelf and then to the top shelf. Participants repeat the task five times and are instructed to perform the task as quickly as possible. The test will be administered for both upper extremities. Test duration is recorded in seconds.
Mortality risk and average life expectancy estimate | one day
  Mortality risk and average life expectancy estimates will be calculated using the Seattle Heart Failure Model. The Seattle Heart Failure Model will be used via the website. The Seattle Heart Failure Model provides consistent 1, 2, and 3 year survival estimates and average life expectancy estimates based on clinical, pharmacological, laboratory, and device information.

SECONDARY OUTCOMES:
functional level | one day
  The New York Heart Association (NYHA) functional classification levels will be determined. NYHA classifies heart patients clinically from 1 to 4 based on their functional status. It is a strong prognostic indicator and risk factor.
hand grip strength | one day
  Hand grip strength will be assessed using a digital hand dynamometer. During the test, patients will be positioned with their arms alongside their bodies, elbows flexed at 90 degrees, and forearms and wrists in a neutral position. Patients will be asked to grasp the fixed dynamometer with maximum force.
upper extremity functional status | one day
  The functional status of the upper extremity will be assessed using the Quick Disability of the Arm, Shoulder, and Hand Questionnaire. Scoring is performed using a 5-point Likert scale. According to this scale, upper extremity activities are scored as follows: 1 no difficulty, 2 mild difficulty, 3 moderate difficulty, 4 severe difficulty, 5 inability to perform. The total score ranges from 0 to 100. "0" indicates that the functions are not affected at all, while "100" indicates that the functions are maximally affected.
lower extremity functional capacity | one day
  Lower extremity functional capacity will be assessed using the one-minute sit-to-stand test. Patients will sit on a back-supported chair without armrests at the start of the test and cross their arms over their shoulders. Starting from this position, patients will be asked to sit down and stand up as quickly as possible for 1 minute. The number of times they sit down and stand up during this 1 minute will be recorded as the test result.
lower extremity performance | one day
  Lower extremity performance will be assessed using a 4-meter walking test. The patient is instructed to start walking at a normal pace on a flat surface measuring 4 meters and to stop at the end of 4 meters. This time is recorded in seconds using a stopwatch.
daily living activities | one day
  Daily living activities will be assessed using the Katz Activities of Daily Living (ADL) Scale. This scale consists of 6 categories: washing, dressing, toileting, transfer, continence, and feeding. Individuals are assessed as follows: 3 points if they can perform daily living activities independently, 2 points if they require partial assistance, and 1 point if they cannot perform the activity at all. In the activities of daily living index, 0-6 points are considered "dependent," 7-12 points are considered "partially dependent," and 13-18 points are considered "independent."
QoL | one day
  Quality of life will be assessed using the Minnesota Quality of Life Scale. This survey consists of 21 questions and asks respondents to answer based on their general situation over the past 4 weeks; it allows for numerical expression ranging from 0 to 5. The total score for this scale is 105. High values indicate low quality of life.
comorbidity | one day
  Comorbidity will be assessed using the Charlson Comorbidity Index. This index includes 19 different diseases rated from 1 to 6, with each disease represented by a specific score. A high CKI Score indicates the presence of additional health problems in the patient and the severity of these problems.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University Faculty of Physical Therapy and Rehabilitation, Ankara, Samanpazarı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided